CLINICAL TRIAL: NCT04185779
Title: COLO-COHORT (Colorectal Cancer Cohort) Study
Status: Recruiting | Type: Observational
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2019-05-29; First posted 2019-12-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Colorectal Neoplasm; Predictive Cancer Model; Model
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA extraction from blood, saliva and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (Cross-sectional arm): This group will comprise of 10,000 patients who have been referred for a colonoscopy. We will be collecting information on their past medical history, smoking history, alcohol history, medication history and family history in addition to their colonoscopy findings. In 6000 of these patients, they will have blood tests, Faecal Immunochemical Test (FIT) level, blood or saliva for DNA extraction and stool microbiome taken. In 4000 of these patients, we will record recent blood tests of interest and they will have no new samples taken. All 10000 patients will also either complete a food frequency questionnaire or endoscopy patient experience questionnaire.
  Interventions: Diagnostic Test: Colonoscopy
- COLO-SPEED (Group B, consent for contact arm): This will be 10,000 patients who will consent for future contact for future research studies.
  Interventions: Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Diagnostic colonoscopy

SUMMARY:
This is a cross-sectional study aimed at identifying factors which best predicts patients at high risk of colorectal cancer or colorectal adenomas and to develop a risk prediction model.

DETAILED DESCRIPTION:
Bowel cancer is the second commonest cause of cancer death in the UK with 16000 people dying per year. Although the NHS Bowel Cancer Screening Programme (BCSP) detects cancers at an earlier stage only 10% of all cancers are detected through screening.

Currently, the only criteria for screening is age and no account is taken of other known risk factors such as smoking, alcohol, family history or obesity. Stool FIT (a new stool test which detects blood that can't be seen with the naked eye) will be introduced into the English BCSP, but there is poor evidence for its use in patients presenting with symptoms. There is also emerging data that there may be differences in the gut bacteria of people with and without cancer or pre cancerous bowel polyps (adenomas).

This will be a national multi-centre study over 5-years. 10000 Patients undergoing colonoscopy as part of BCSP or due to symptoms will be recruited. Patients will be asked to fill in a health questionnaire, have their height, weight, waist circumference measured. Patients will also receive blood tests, stool tests or saliva tests depending on the indication for their colonoscopy. The results of the colonoscopy and any samples taken will be collated. Patients will receive a patient experience questionnaire or food frequency questionnaire. A further 10,000 patients from the North of England will be consented to be contacted for future studies with some of the information above collected.

The aim of this study is to develop a risk prediction model to help determine which patients are at highest risk of having adenomas or bowel cancer. The investigators will also explore the significance of the gut bacteria composition in patients with adenomas or cancer to help inform this risk model. Additionally the investigators will develop a large platform of patients who consent to be contacted for future research.

ELIGIBILITY:
Inclusion Criteria:

Group A

* Aged ≥30 years* and able to give informed consent
* Patients attending colonoscopy

  * Through Bowel Cancer Screening Programme (FIT positive, Bowelscope conversion, surveillance)
  * Through standard NHS care (most commonly due to iron deficiency anaemia, altered bowel habit, weight loss, rectal bleeding, planned polypectomy**, those referred on basis of family history, abnormal cross-sectional imaging, polyp surveillance or post CRC surveillance)

    * The age of 30 was chosen to ensure that this is a population likely to be enriched for colorectal neoplasia with neoplasia below this age uncommon **In those attending for planned polypectomy, the results from the initial colonoscopy and the endoscopy where the polypectomy is undertaken will be summated for purposes of calculating the neoplasia profile

(COLO-SPEED) Group B

* Any patient attending for colonoscopy and able to give informed consent
* ≥ 18 years old
* Patient from the North of England

Exclusion Criteria:

Group A

* Unable to give informed consent
* Known polyposis syndrome
* Previous total colectomy
* Known colonic stricture which would limit complete colonoscopy
* Attending for planned therapeutic procedure other than polypectomy, such as insertion of colonic stent
* Attending for assessment of known inflammatory bowel disease (IBD) activity or for IBD surveillance
* Patients currently recruited into an interventional CTIMP for CRC prevention*

COLO-SPEED (Group B) **

* Unable to give informed consent
* Not in a centre supported by COLO-SPEED infrastructure (North of England)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred for a colonoscopy (minimum age limits as above in inclusion criteria) either through the bowel cancer screening programme, as part of a surveillance programme or due to symptoms
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of colorectal neoplasia | 5 years
  Incidence of colorectal neoplasia (colorectal cancer and advanced adenomas)

SECONDARY OUTCOMES:
Stool microbiome pattern | 5 years
  Assessing trends in variation of stool microbiome in patients with normal colon, adenomas, bowel cancer)
Number of participants who consent for future contact | 5 years
  A registry of patients who consent to be contacted in the future for future research studies

CONTACTS AND LOCATIONS:
Overall Officials: Colin Rees, Principal Investigator — Newcastle University
Locations (3):
- United Kingdom (3):
  - South Tyneside and Sunderland NHS Foundation Trust, South Shields, Tyne and Wear
  - Kettering General Hospitals NHS Foundation Trust, Kettering
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No